CLINICAL TRIAL: NCT00757406
Title: Assessment of Unilateral Lymphoedema of the Leg
Status: Completed | Type: Observational
Sponsor: ImpediMed Limited (Industry)
Responsible Party: Dr Robyn Box, Queensland Lymphoedema and Breast Oncology Physiotherapy
Other Study IDs: UQLDEX02
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Lymphedema
Keywords: Lymphedema; Bioimpedance
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Test group - Lymphedema sufferers
- 2: Control group - healthy volunteers

SUMMARY:
To demonstrate that ImpediMed L-Dex U400 can be used to assess unilateral Lymphoedema of the leg using the same principles for arms.

DETAILED DESCRIPTION:
When Lymphoedema is present, lymph and other fluids build up in the interstitial spaces of the tissues. This results in an overall increase in the total amount of extracellular fluid (ECF) in the limb, causing swelling. This can be documented by measuring the impedance (opposition) to a low frequency current that has been passed into the limb. Low frequency current travels predominantly through the ECF, where the Lymphoedema manifests. As the fluid builds up in the limb, the impedance to the current decreases and it is in this way that low frequency bioimpedance is able to assess Lymphoedema.

Multi-frequency bio-impedance analysis otherwise known as Bioimpedance Spectroscopy (BIS) has been reported to be effective for the measurement of ECF and sub clinical changes in ECF to predict the onset of Lymphoedema in the arms in studies conducted by Cornish et al. It has been reported by Warren et al that BIS can be used as a reliable and accurate tool for documenting presence of lymphoedema in patients with wither upper- or lower-extremity swelling.

The L-Dex U400 device uses an "impedance ratio" methodology to assess unilateral Lymphoedema of the arm. By this method the unaffected arm acts as an internal and subject specific control. The strategy of this study is to show that the L-Dex U400 can use this methodology to assess unilateral leg Lymphoedema.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Be between the ages of 18-75 years.
* Self-describe general health as satisfactory.
* Understand the proposed study and be willing and fully able to comply with the study procedures.
* Be a willing participant and be capable of giving and has given informed written consent for entry into the study.
* Have been previously diagnosed, by current clinical practice, as having unilateral Lymphoedema of the leg.

Group 2:

* Be between the ages of 18-75 years.
* Self-describe general health as satisfactory.
* Understand the proposed study and be willing and fully able to comply with the study procedures.
* Be a willing participant and be capable of giving and has given informed written consent for entry into the study.

Exclusion Criteria:

* Have a known heart condition or an implantable device such as a pacemaker or ICD.
* Have a metallic surgical implant (e.g. total hip replacement) not including small implants such as sternal wires or surgical staples.
* Suffer from a renal disorder.
* Be taking diuretic medications.
* Have consumed large amounts of alcohol or caffeinated beverages within six hours of the study.
* Have undertaken excessive exercise within two hours of BIA
* Have a reported fever of > 38°C at time of screening.
* Be currently in the fourth week of the menstrual cycle.
* Be pregnant or currently breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 - Test group - will be recruited through advertisements placed at Qld Lymphoedema and Breast Oncology Physiotherapy, Lymphoedema Association of QLD, Gynecological Cancer Support Group and notification to other private therapists to inform them of the study.
  Group 2 - Control group - will be through advertisements placed at Qld Lymphoedema and Breast Oncology Physiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
That the L-Dex U400 detects Unilateral leg lymphedema in subjects with the condition and does not detect it in subjects without the condition. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robyn C Box, PhD, Principal Investigator — Qld Lymphoedema and Breast Oncology Physiotherapy
Locations (1):
- Qld Lymphoedema and Breast Oncology Physiotherapy, Brisbane, Queensland, Australia